CLINICAL TRIAL: NCT07284459
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Oral PIPE 791 in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of PIPE 791 in Subjects With Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Contineum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTX-791-201
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; PIPE 791; Pulmonary Fibrosis; IPF; ILD; Interstitial lung disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PIPE-791 Dose A (Experimental)
  Interventions: Drug: PIPE-791 Dose A
- PIPE-791 Dose B (Experimental)
  Interventions: Drug: PIPE-791 Dose B
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PIPE-791 Dose A — Subjects will receive a daily oral dose of PIPE-791 in tablet form
  Other Names: PIPE-791
  Arms: PIPE-791 Dose A
Drug: PIPE-791 Dose B — Subjects will receive a daily oral dose of PIPE-791 in tablet form
  Other Names: PIPE-791
  Arms: PIPE-791 Dose B
Drug: Placebo — Subjects will receive a daily oral dose of matching Placebo in tablet form
  Arms: Placebo

SUMMARY:
This is a Ph 2, randomized, double-blind, placebo-controlled global multicenter study to evaluate the efficacy, safety, tolerability, and pharmacokinetics (PK) of PIPE-791 in subjects with a diagnosis of Idiopathic Pulmonary Fibrosis (IPF) with or without background treatment.

DETAILED DESCRIPTION:
This is a Ph 2, randomized, double-blind, placebo-controlled global multicenter study to evaluate the efficacy, safety, tolerability, and PK of PIPE-791 in subjects with a diagnosis of Idiopathic Pulmonary Fibrosis with or without background treatment. The treatment period is 26 weeks and full study duration is up to 36 weeks including Screening and Follow-Up. Approximately 324 subjects will be enrolled into one of three treatment arms, PIPE-791 Dose A, PIPE-791 Dose B, or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥ 40 years of age at the time of Randomization
* A diagnosis of IPF within 7 years prior to Screening, based on the 2018 ATS/ERS/JRS/ALAT practice guideline as confirmed by the Investigator, and a centrally read screening HRCT with verification of usual interstitial pneumonia
* Percent predicted (pp) FVC ≥ 40% on Screening spirometry
* Subjects may enter the study whether or not they are receiving background antifibrotic therapy, approved for the treatment of IPF (nintedanib or pirfenidone, but not both concurrently)

Key Exclusion Criteria:

* Those with a history of interstitial lung disease (ILD) other than IPF are not eligible.
* Those with pulmonary arterial hypertension (PAH) requiring multi-drug therapy are not eligible.
* Those who have experienced an IPF exacerbation within 6 weeks of Screening, or during Screening, are not eligible.
* Those with an estimated glomerular filtration rate (eGFR) ≤ 30 ml/min/1.73 m2 (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) (Inker 2021) or who have Child-Pugh Class B or C hepatic impairment are not eligible.

Additional inclusion and exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Absolute change in forced vital capacity (FVC) (mL) | From baseline to Week 26

SECONDARY OUTCOMES:
To investigate the safety and tolerability of PIPE-791 compared to placebo based on percentage of treatment-emergent adverse events (TEAE) | From baseline to Week 30
Relative change in FVC (mL) | From baseline to Week 26
  Additional assessment of disease progression through lung function measurements
Proportion of subjects with a ≥10% absolute decline in percent predicted FVC (ppFVC) | From baseline to Weeks 12 and Week 26
Time to first ≥10% absolute decline in ppFVC | From baseline to time of first ≥10% absolute decline, up to Week 26
Absolute change in ppFVC | From baseline to Week 26
  Additional assessment of disease progression through lung function measurements
Relative change in ppFVC | From baseline to Week 26
  Additional assessment of disease progression through lung function measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mudiaga O Sowho, MD, MPH, Study Director — Contineum Therapeutics
Locations (2):
- Canada (2):
  - Dynamic Drug Advancement Ltd., Ajax, Ontario
  - Dr. Anil Dhar Medicine Professional Corporation, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No